CLINICAL TRIAL: NCT04786730
Title: A Phase 1b, Multicenter, Open-label, Multiple Ascending Dose Trial to Assess the Pharmacokinetics, Safety, and Tolerability of Centanafadine Extended-release Capsules After Oral Administration in Pediatric Subjects (4 to 12 Years, Inclusive) With Attention-deficit Hyperactivity Disorder
Brief Title: A Trial to Assess the Pharmacokinetics, Safety, and Tolerability of Centanafadine Capsules in Pediatric Subjects With Attention-deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 405-201-00046
Record Dates: First submitted 2021-02-25; First posted 2021-03-08 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Attention-deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label centanafadine (Experimental): There will be multiple cohorts dosed with open-label centanafadine.
  Interventions: Drug: Centanafadine

INTERVENTIONS:
Drug: Centanafadine — Doses of centanafadine will be taken once daily in the morning on Days 1 through 14. The fixed dose strengths will be administered according to body weight. Up to 12 subjects will be enrolled in the 9 to 12 years age cohorts (Cohorts 1 and 6), up to 8 subjects will be enrolled in each of the 6 to 8 years age cohorts (Cohorts 2 and 3), and up to 5 subjects will be enrolled in each of the 4 to 5 years age cohorts (Cohorts 4 and 5).

SUMMARY:
This is a phase 1b, multicenter, open-label, multiple-dose trial in pediatric subjects (4 - 12 years of age, inclusive) with a confirmed diagnosis of ADHD.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects 4 to 12 years of age, inclusive, at the time of informed consent/assent.
* A diagnosis of any ADHD subtype based on Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5) criteria and confirmed by the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).

Key Exclusion Criteria:

* Subjects with a clinical presentation or history that is consistent with delirium, dementia, amnesia, or other cognitive disorders; subjects with psychiatric symptoms that are better accounted for by another general medical condition(s) or direct effect of a substance (medication, illicit drug use, etc); or subjects with a clinical presentation or history of psychotic symptoms.
* Subjects with developmental disorders, such as autism spectrum disorder.
* Subjects with a history of intellectual disability as determined by at least 1 of the following: intelligence quotient < 70, or clinical evidence, or a social or school history that is suggestive of intellectual disability.
* Subjects who currently have clinically significant neurological, dermatological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders such as any history of myocardial infarction, congestive heart failure, HIV seropositive status/ AIDS, or chronic hepatitis B or C.
* Subjects who have history of clinically significant tachycardia or hypertension.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Maximal peak plasma concentration (Cmax) | 24 hours
Area under the concentration-time curve from time 0 to 24 hours (AUC0-24h) on day 14 | 24 hours
Apparent clearance and apparent volume of distribution of centanafadine on Day 14 | 24 hours

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - For additional information regarding sites, contact 844-687-8522, Little Rock, Arkansas
  - For additional information regarding sites, contact 844-687-8522, Decatur, Georgia
  - For additional information regarding sites, contact 844-687-8522, Las Vegas, Nevada
  - For additional information regarding sites, contact 844-687-8522, Oklahoma City, Oklahoma
  - For additional information regarding sites, contact 844-687-8522, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: http://clinical-trials.otsuka.com